CLINICAL TRIAL: NCT02892903
Title: A Randomised Controlled Trial to Compare Routine Pressure Wire Assessment With Conventional Angiography in the Management of Patients With Coronary Artery Disease.
Brief Title: In the Management of Coronary Artery Disease, Does Routine Pressure Wire Assessment at the Time of Coronary Angiography Affect Management Strategy, Hospital Costs and Outcomes?
Acronym: RIPCORD 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RHM CAR0498
Record Dates: First submitted 2016-07-06; First posted 2016-09-08 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Chest Pain; Stable Angina; Acute Coronary Syndrome; Non ST Segment Elevation Acute Coronary Syndrome
Keywords: Fractional flow reserve (FFR); Pressure wire (PW); Coronary angiography
MeSH Terms: conditions — Chest Pain; Angina, Stable; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional angiography (No Intervention): Routine angiography will be performed according to local best practice
- Routine Measurement of FFR (Experimental): Additional investigation with the measurement of FFR in all major vessels
  Interventions: Device: Routine Measurement of FFR

INTERVENTIONS:
Device: Routine Measurement of FFR — FFR measurement will be performed in all major vessels with normal (TIMI 3) flow. Occluded vessels and vessels with TIMI flow <3 will not be examined but will be 'awarded' an FFR value of 0.5
  Other Names: Pressure wire assessment
  Arms: Routine Measurement of FFR

SUMMARY:
A randomised controlled trial to compare two strategies for the investigation of coronary artery disease at the time of angiography. Patients will be randomised to conventional angiography or additional, routine pressure wire assessment - measuring fractional flow reserve (FFR) - in all main vessels judged as being of sufficient vessel calibre to allow percutaneous coronary intervention (PCI) (experimental arm).

DETAILED DESCRIPTION:
The study will recruit patients undergoing angiography for the investigation of stable angina or for the assessment of a recent, but stabilised, non-ST elevation acute coronary syndrome event. Eligible patients who provide written informed consent will be randomised to conventional angiography or additional, routine pressure wire assessment - measuring fractional flow reserve (FFR) - in all main vessels judged as being of sufficient vessel calibre to allow percutaneous coronary intervention (PCI) (experimental arm). The study pragmatic design allows investigators to conduct all diagnostic and therapeutic management in accordance with prevailing best practice patterns. Study outcome measures will examine resource utilisation, patient reported quality of life and clinical events at 1 year.

ELIGIBILITY:
· Inclusion criteria

o Outline Initial Inclusion Criteria (before entry to cath lab):

Patient scheduled for coronary angiography for the:

* Elective investigation of known or suspected coronary artery disease OR
* Urgent investigation of a recent but stabilised, non-ST elevation acute coronary syndrome event

  o Outline Angiographic Inclusion Criterion (after angiography):
* Presence of significant coronary disease defined as:

Any stenosis >30% reduction in luminal diameter, by visual estimate, in at least one vessel (main or branch) of sufficient calibre to permit the potential performance of PCI - approximately 2.25 mm diameter.

* Key Exclusion Criteria

  * Screening phase exclusion criteria:

    * ≤ 18 years of age
    * Previous enrolment in this trial
    * Currently enrolled into another study unless co-enrolment approved by Chief Investigator (CI) and the clinical trials unit (CTU)
    * Inability to provide informed consent
    * Residence outside the United Kingdom (UK) or other issues limiting the ability to secure clinical follow-up data to one year
    * Non-cardiac pathology that may limit survival in the next year
    * Clear contraindication to potential future management with CABG or PCI (patients should be a potential candidate for medical therapy or revascularisation with either PCI or surgery)
    * Heart valve disease of sufficient import to consider valve replacement or other intervention as part of an index management strategy
    * Hypertrophic cardiomyopathy
    * Previous coronary artery surgery of any type
    * Known chronic renal impairment with a current estimated glomerular filtration rate (eGFR) of < 45
    * Anaemia with a current measured haemoglobin of < 100
    * Angiography performed in the context of an ST elevation myocardial infarction event
    * Any patient who at the time of planned angiography manifests haemodynamic instability, or recurrent sustained ventricular arrhythmia, or Mobitz type II or complete heart block
    * Any patient who at the time of planned angiography manifests unstable chest pain symptoms at rest or has required the continuing use of intravenous nitrates or regular opioid analgesia to control symptoms
    * Continuing use of intravenous glycoprotein 2b/3a (GP2b3a) agents before entry to the catheterisation laboratory
    * Known intolerance, hypersensitivity or contraindication to adenosine - including significant reversible airways disease
    * Additional investigations planned (or deemed likely to be required) for the assessment of myocardial ischaemia or viability. Examples of proposed tests that would constitute an exclusion criterion would include, but are not limited to, exercise tolerance testing, stress echocardiography, cardiac MRI viability or perfusion scanning or nuclear myocardial perfusion scanning.
    * Active bleeding at the time of planned index angiography
    * Pregnant women
  * Angiographic phase exclusion criteria:

    * Single vessel occlusive coronary disease (TIMI flow <3) as sole disease
    * Patient not suitable for the immediate performance of a pressure wire assessment of all major vessels for any reason, for example:

      * Patient discomfort
      * Change in the clinical condition or complication of angiography requiring termination of the procedure or immediate intervention
      * Significant use of radiographic contrast or X-Ray exposure during the initial angiography
      * Inadequate angiographic images or failure to intubate any of the coronary vessels
      * Aorto-ostial disease that would preclude accurate assessment of FFR
      * Insufficient laboratory time
      * Uncertain availability of key clinical and trial staff
      * PW use in coronaries declared unsafe (e.g. tight or long disease)
      * PW use in coronaries declared unsuitable (e.g. distal disease or complete cross-filling)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Primary Economic Outcome Measure | One year
  Resource utilisation as determined by hospital care costs at one year; All hospital admissions will be tracked using national hospital episode statistics; the cost of each episode will be derived from a cost model using standard UK tariffs. This analysis will compare the mean (or median) of the total hospital costs recorded for each patient over the 12 month follow-up period.
Primary Quality of Life Outcome Measure | One year
  Patient reported quality of life at one year using the EQ-5D health questionnaire.

SECONDARY OUTCOMES:
Management strategy information | Reported once: Single declaration at index procedure after randomisation
  · Proportion of vessels deemed to demonstrate flow-limiting disease and targeted for revascularisation in the declared initial management strategy.
Management strategy information | Reported once: Single declaration at index procedure after randomisation
  · Proportion of patients scheduled for management with medical therapy, percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) in the declared initial management strategy.
Angina symptoms | One year
  • Angina symptoms as reported by the research team after the 12 month contact, described by Canadian Cardiovascular Society Grade.
Angina symptoms | One year
  • Angina symptoms as reported by the patient with private completion of a screening form at 12 months, described by Canadian Cardiovascular Society Grade.
All-cause mortality | One year
Number of hospitalisation events | One year
Total hospital days | One year
Hospitalisation events | One year
  Hospitalisation events coded as cerebro-vascular accident (CVA).
Hospitalisation events | One year
  Hospitalisation events coded as myocardial infarction.
Hospitalisation events | One year
  Hospitalisation events coded as Coronary revascularisation. This analysis will involve a pre-specified subgroup analysis of:
  * Planned revascularisation - if declared as the index strategy.
  * All additional revascularisation events.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Curzen, BM PhD FRCP, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Rod H Stables, MA, DM, BM BCH, FRCP, Principal Investigator — Liverpool Heart and Chest Hospital NHS Foundation Trust
Locations (17):
- United Kingdom (17):
  - Royal Bournemouth Hospital - The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth, Dorset
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Queen Alexandra Hospital - Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire
  - Southampton General Hospital - University Hospitals Southampton NHS Foundation Trust, Southampton, Hampshire
  - Royal Blackburn Teaching Hospital - East Lancashire Hospitals NHS Trust, Blackburn, Lancashire
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, Merseyside
  - Freeman Hospital - Newcastle Hospitals, Newcastle upon Tyne, Northumberland
  - King's Mill Hospital - Sherwood Forest Hospitals NHS Foundation Trust, Mansfield, Nottinghamshire
  - City Hospital - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Golden Jubilee National Hospital, Glasgow, Scotland
  - Northern General Hospital - Sheffield Teaching Hospitals, Sheffield, South Yorkshire
  - Royal Stoke University Hospital - University Hospitals of North Midlands, Stoke-on-Trent, Staffordshire
  - Queen Elizabeth Hospital - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Pinderfields Hospital - The Mid Yorkshire Hospitals NHS Trust, Wakefield, West Yorkshire
  - Castle Hill Hospital - Hull and East Yorkshire Hospitals NHS Trust, Hull, Yorkshire
  - Leeds General Infirmary - Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire
  - Bristol Heart Institute - University Hospitals Bristol NHS Foundation Trust, Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zir LM, Miller SW, Dinsmore RE, Gilbert JP, Harthorne JW. Interobserver variability in coronary angiography. Circulation. 1976 Apr;53(4):627-32. doi: 10.1161/01.cir.53.4.627. PMID 1253383
- [Background] White CW, Wright CB, Doty DB, Hiratza LF, Eastham CL, Harrison DG, Marcus ML. Does visual interpretation of the coronary arteriogram predict the physiologic importance of a coronary stenosis? N Engl J Med. 1984 Mar 29;310(13):819-24. doi: 10.1056/NEJM198403293101304. PMID 6700670
- [Background] De Bruyne B, Baudhuin T, Melin JA, Pijls NH, Sys SU, Bol A, Paulus WJ, Heyndrickx GR, Wijns W. Coronary flow reserve calculated from pressure measurements in humans. Validation with positron emission tomography. Circulation. 1994 Mar;89(3):1013-22. doi: 10.1161/01.cir.89.3.1013. PMID 8124786
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Berger A, Botman KJ, MacCarthy PA, Wijns W, Bartunek J, Heyndrickx GR, Pijls NH, De Bruyne B. Long-term clinical outcome after fractional flow reserve-guided percutaneous coronary intervention in patients with multivessel disease. J Am Coll Cardiol. 2005 Aug 2;46(3):438-42. doi: 10.1016/j.jacc.2005.04.041. PMID 16053955
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Background] Pijls NH, Fearon WF, Tonino PA, Siebert U, Ikeno F, Bornschein B, van't Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, De Bruyne B; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention in patients with multivessel coronary artery disease: 2-year follow-up of the FAME (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation) study. J Am Coll Cardiol. 2010 Jul 13;56(3):177-84. doi: 10.1016/j.jacc.2010.04.012. Epub 2010 May 28. PMID 20537493
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Longman K, Curzen N. Should ischemia be the main target in selecting a percutaneous coronary intervention strategy? Expert Rev Cardiovasc Ther. 2013 Aug;11(8):1051-9. doi: 10.1586/14779072.2013.814856. PMID 23984928
- [Background] Toth G, Hamilos M, Pyxaras S, Mangiacapra F, Nelis O, De Vroey F, Di Serafino L, Muller O, Van Mieghem C, Wyffels E, Heyndrickx GR, Bartunek J, Vanderheyden M, Barbato E, Wijns W, De Bruyne B. Evolving concepts of angiogram: fractional flow reserve discordances in 4000 coronary stenoses. Eur Heart J. 2014 Oct 21;35(40):2831-8. doi: 10.1093/eurheartj/ehu094. Epub 2014 Mar 18. PMID 24644308
- [Background] Curzen N, Rana O, Nicholas Z, Golledge P, Zaman A, Oldroyd K, Hanratty C, Banning A, Wheatcroft S, Hobson A, Chitkara K, Hildick-Smith D, McKenzie D, Calver A, Dimitrov BD, Corbett S. Does routine pressure wire assessment influence management strategy at coronary angiography for diagnosis of chest pain?: the RIPCORD study. Circ Cardiovasc Interv. 2014 Apr;7(2):248-55. doi: 10.1161/CIRCINTERVENTIONS.113.000978. Epub 2014 Mar 18. PMID 24642999
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on behalf of the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction. Third universal definition of myocardial infarction. Glob Heart. 2012 Dec;7(4):275-95. doi: 10.1016/j.gheart.2012.08.001. Epub 2012 Sep 26. No abstract available. PMID 25689940
- [Background] Weintraub WS, Mahoney EM, Zhang Z, Chu H, Hutton J, Buxton M, Booth J, Nugara F, Stables RH, Dooley P, Collinson J, Stuteville M, Delahunty N, Wright A, Flather MD, De Cock E. One year comparison of costs of coronary surgery versus percutaneous coronary intervention in the stent or surgery trial. Heart. 2004 Jul;90(7):782-8. doi: 10.1136/hrt.2003.015057. PMID 15201249
- [Background] Zhang Z, Mahoney EM, Stables RH, Booth J, Nugara F, Spertus JA, Weintraub WS. Disease-specific health status after stent-assisted percutaneous coronary intervention and coronary artery bypass surgery: one-year results from the Stent or Surgery trial. Circulation. 2003 Oct 7;108(14):1694-700. doi: 10.1161/01.CIR.0000087600.83707.FD. Epub 2003 Sep 15. PMID 12975252
- [Background] SoS Investigators. Coronary artery bypass surgery versus percutaneous coronary intervention with stent implantation in patients with multivessel coronary artery disease (the Stent or Surgery trial): a randomised controlled trial. Lancet. 2002 Sep 28;360(9338):965-70. doi: 10.1016/S0140-6736(02)11078-6. PMID 12383664
- [Background] Van Belle E, Rioufol G, Pouillot C, Cuisset T, Bougrini K, Teiger E, Champagne S, Belle L, Barreau D, Hanssen M, Besnard C, Dauphin R, Dallongeville J, El Hahi Y, Sideris G, Bretelle C, Lhoest N, Barnay P, Leborgne L, Dupouy P; Investigators of the Registre Francais de la FFR-R3F. Outcome impact of coronary revascularization strategy reclassification with fractional flow reserve at time of diagnostic angiography: insights from a large French multicenter fractional flow reserve registry. Circulation. 2014 Jan 14;129(2):173-85. doi: 10.1161/CIRCULATIONAHA.113.006646. Epub 2013 Nov 19. PMID 24255062
- [Background] Henderson R, Lee L. The epidemiology and pathophysiology of coronary artery disease. Chapter 1 in The Oxford Textbook of Interventional Cardiology. Eds: Redwood, Curzen, Thomas. Oxford University Press 2010.
- [Background] Muller O, De Bruyne B. Coronary physiology in clinical practice. Chapter 9 in in The Oxford Book of Interventional Cardiology. Eds: Redwood, Curzen, Thomas. Oxford University Press 2010.
- [Background] Chest Pain of Recent Onset. NICE Guidance CG95, 2010. https://www.nice.org.uk/guidance/CG95
- [Derived] Elguindy M, Stables R, Nicholas Z, Kemp I, Curzen N. Design and Rationale of the RIPCORD 2 Trial (Does Routine Pressure Wire Assessment Influence Management Strategy at Coronary Angiography for Diagnosis of Chest Pain?): A Randomized Controlled Trial to Compare Routine Pressure Wire Assessment With Conventional Angiography in the Management of Patients With Coronary Artery Disease. Circ Cardiovasc Qual Outcomes. 2018 Feb;11(2):e004191. doi: 10.1161/CIRCOUTCOMES.117.004191. PMID 29449442